CLINICAL TRIAL: NCT04411836
Title: Effectiveness of Novel Approaches to Radical Cure With Tafenoquine and Primaquine - a Randomized Controlled Trial in P. Vivax Patients
Brief Title: Effectiveness of Novel Approaches to Radical Cure With Tafenoquine and Primaquine
Acronym: EFFORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: University of Melbourne (Other); National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); Mahidol Oxford Tropical Medicine Research Unit (Other); Ethiopian Public Health Institute (Other Government); Universitas Sumatera Utara (Other); Arba Minch University (Other); Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFORT
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Vivax Malaria; Plasmodium Vivax; Malaria, Vivax; Malaria Relapse
Keywords: tafenoquine; primaquine
MeSH Terms: conditions — Malaria, Vivax | interventions — tafenoquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): Patients are treated with schizontocidal treatment plus low dose PQ (total dose 3.5mg/kg) unsupervised over 14 days (PQ14)
- PQ Intervention (Experimental): Patients are treated with schizontocidal treatment plus high dose PQ (total dose 7 mg/kg) unsupervised over 7 days (PQ7)
  Interventions: Drug: Primaquine
- TQ Intervention (Experimental): Patients are treated with schizontocidal treatment plus a single dose of Tafenoquine (TQ)
  Interventions: Drug: Tafenoquine

INTERVENTIONS:
Drug: Tafenoquine — patients are treated with schizontocidal treatment plus a single dose of Tafenoquine (TQ).
  Arms: TQ Intervention
Drug: Primaquine — patients are treated with schizontocidal treatment plus high dose PQ (total dose 7 mg/kg) unsupervised over 7 days (PQ7)
  Other Names: Primaquine 7 days
  Arms: PQ Intervention

SUMMARY:
Health care facility based, randomized, controlled, open label, superiority trial with 3 arms

DETAILED DESCRIPTION:
* To assess the effectiveness of a short-course of high dose primaquine (total dose 7mg/kg given unsupervised over 7 days) compared to the current standard low dose primaquine regimen (total dose 3.5mg/kg given unsupervised over 14 days).
* To assess the effectiveness of tafenoquine (single dose of 300mg) compared to the short-course high dose primaquine regimen.
* To assess the safety of tafenoquine compared to the high and low dose primaquine regimens.
* To assess the cost-effectiveness and feasibility of high dose primaquine and tafenoquine compared to the current low dose primaquine regimen

ELIGIBILITY:
Inclusion Criteria

* P. vivax peripheral parasitaemia (mono-infection) as determined by microscopy
* G6PD normal status (G6PD activity ≥ 70% of the adjusted male median as determined by the Biosensor™ (SD Biosensor, ROK))
* Fever (temperature ≥37.5⁰C) or history of fever in the preceding 48 hours
* Age ≥18 years
* Written informed consent
* Living in the study area and willing to be followed for six months

Exclusion Criteria:

* Danger signs or symptoms of severe malaria
* Anaemia (defined as Hb <8g/dl)
* Pregnant or lactating females
* Known hypersensitivity to any of the study drugs
* Regular use of drugs with haemolytic potential

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence risk any P vivax PQ7 / PQ14 | 6 months
  The incidence risk (time to first event) of any P. vivax parasitaemia during the 6-month follow up period as determined by microscopy compared between the PQ7 arm and the control arm (PQ14).

SECONDARY OUTCOMES:
Incidence risk any P vivax PQ7 / TQ | 6 months
  The incidence risk (time to first event) of any P. vivax parasitaemia during the 6 months follow up period as determined by microscopy compared between PQ7 and TQ arms
Incidence risk symptomatic P vivax TQ / PQ14 | 6 months
  The incidence risk (time to first event) of symptomatic P. vivax parasitaemia during the 6 months follow up period as determined by microscopy compared between TQ and the control arm (PQ14).
Incidence risk any P vivax PQ7 / PQ14 | 6 months
  The incidence risk (time to first event) of symptomatic P. vivax parasitaemia during the 6-month follow up period as determined by microscopy compared between the PQ7 arm and the control arm (PQ14).
Incidence risk any P vivax PQ7 / TQ | 6 months
  • The incidence risk (time to first event) of any P. vivax parasitaemia during the 6 months follow up period as determined by microscopy compared between PQ7 and TQ arms
Incidence risk any P vivax PQ14 / TQ | 6 months
  The incidence risk (time to first event) of any P. vivax parasitaemia during the 6 months follow up period as determined by microscopy compared between PQ14 and TQ arms

CONTACTS AND LOCATIONS:
Overall Officials: Kamala Thriemer, MD, MPH, PhD, Principal Investigator — Menzies School of Health Research
Locations (6):
- Cambodia (3):
  - Kravanh District Hospital, Pursat, Pursat
  - Chambak Health Center, Kampong Speu
  - Siem Pang Health Centre, Stung Treng
- Arba Minch General Hospital, Arba Minch, Ethiopia
- Tanjung Leidong Health Center, Labuhanbatu, Sumatera, Indonesia
- Aga Khan Hospital Karachi, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be made available to others. Data collected for the study, including individual patient data and the final trial dataset are reserved for the chief investigator and co-investigators of the trial. The trial will be reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines. Trial results will be published in peer-reviewed open access journals and disseminated to trial stakeholders, including participants, as per ethical guidelines.
Supporting Information: Study Protocol, SAP
Access Criteria: The data are available for access via the WorldWide Antimalarial Resistance Network (WWARN.org). Requests for access will be reviewed by a Data Access Committee to ensure that use of data protects the interests of the participants and researchers according to the terms of ethics approval and principles of equitable data sharing. Requests can be submitted by email to malariaDAC@iddo.org via the Data Access Form available at WWARN.org/accessing-data. The WWARN is registered with the Registry of Research Data Repositories (re3data.org).
URL: http://WWARN.org/accessing-data